CLINICAL TRIAL: NCT01465178
Title: Improving the Understanding of the Response to Vitamin D Supplementation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2011-0601
Record Dates: First submitted 2011-10-27; First posted 2011-11-04 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Deficiency
Keywords: hypovitaminosis D; vitamin D insufficiency; low vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2000 IU vitamin D3 (Active Comparator): Cholecalciferol 2,000 IU capsules
  Interventions: Dietary Supplement: cholecalciferol
- Placebo (Placebo Comparator): Non-matching placebo, gelatin filled capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 2000 IU cholecalciferol gelcaps by mouth daily
  Arms: 2000 IU vitamin D3
Dietary Supplement: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
It is the investigators hypothesis that the current method of evaluating vitamin D status, measuring circulating 25-hydroxy vitamin D is not providing the full metabolic picture, and is therefore inadequate. The investigators liken this concept to the evolution of cholesterol where initially, total cholesterol was the only measurement, and have since determined the importance of HDL, LDL and triglycerides in evaluating patient status. Similarly, the investigators feel measurement of other vitamin D components such as sulfated vitamin D, circulating vitamin D3 and 3-epi 25-hydroxy vitamin D will offer more comprehensive information about a patient's vitamin D status.

It is our overarching hypothesis that a "vitamin D assay panel," will enhance understanding of vitamin D status. It is our expectation that the enhanced understanding based on improved measurement capability will ultimately translate to improved definition of vitamin D status and need for supplementation on an individual level.

DETAILED DESCRIPTION:
This hypothesis is supported by several observations. First, recent work finds previously unappreciated vitamin D metabolites, notably 3 epi-25(OH)D348 and sulfated 25(OH)D3, in virtually all human sera and circulating in amounts that vary widely between individuals. These compounds may be measured by current "25(OH)D" assays,46, 63 and thereby confound accuracy of such measurements. Secondly, substantial but inadequately understood variability of 25(OH)D response to supplementation and UV exposure exists.15, 42-44 It is likely that currently unappreciated genetic and/or physiologic factors, e.g., differences in absorption or degradation, underpin these observations. Our panel will allow definition of these differences. Finally, the inadequacy of our current approach to classify vitamin D status (singular 25(OH)D measurement) is exemplified by the great between-individual variability in the PTH/25(OH)D relationship as noted above.8, 64 Thus, the investigators believe that exploration of a "vitamin D assay panel," consisting of measurements that reflect input (cholecalciferol and ergocalciferol) and confounders to the 25(OH)D assay [3 epi-25(OH)D and sulfated 25(OH)D] is essential to accurately define optimal vitamin D status and to determine the ideal approach for vitamin D repletion.

To begin testing this hypothesis, the Specific Aims of this research are to document the vitamin D profile response defined as change in serum concentration of:

1. 25(OH)D
2. cholecalciferol
3. 3 epi-25(OH)D
4. Sulfated 25(OH)D following four months of supplementation with 2,200 IU of daily vitamin D3 in postmenopausal women. Our primary outcome variable is the effect of supplementation on serum 25(OH)D3; secondary outcomes are change in cholecalciferol, 3 epi-25(OH)D3 and sulfated 25(OH)D3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, community-dwelling ambulatory postmenopausal White, non-Hispanic women
* Able and willing to sign informed consent
* Baseline serum 25(OH)D concentration of 10-29 ng/mL
* Willing to not alter the amount of their baseline vitamin D supplementation during the course of this study
* Willing to use sunscreen (SPF ≥15) when sun exposure of > 15 minutes is expected

Exclusion Criteria:

* Presence of any measurable circulating 25(OH)D2 on screening measurement
* Current hypercalcemia (serum calcium > 10.5 mg/dl) or untreated primary hyperparathyroidism
* History of nephrolithiasis
* Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis
* History of any form of cancer within the past five years with the exception of adequately treated squamous cell or basal cell skin carcinoma
* Renal failure; defined as a calculated creatinine clearance (using the Cockroft-Gault approach) of ≤ 35 ml/minute
* Severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study
* Known metabolic bone disease, e.g., Paget's disease, osteomalacia
* Treatment with any drug known to interfere with vitamin D metabolism, e.g., phenytoin, phenobarbital
* Treatment with high dose vitamin D (≥ 50,000 IU weekly) or any active metabolites of vitamin D, e.g., calcitriol, within six months of screening
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer
* Planned trips/vacations likely to be associated with substantial amounts of sun exposure during the course of the study

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started December 2011 and ended December 2014. Subjects were enrolled from the community and research was conducted at the University of Wisconsin Osteoporosis Clinical Research Program.
Pre-assignment Details: No adverse events were reported between screening and randomization. All screened volunteers that were not enrolled in the study were deemed ineligible based on 25(OH)vitamin D being outside the study entry criterion.
Period: Overall Study
Arm/Group | 2000 IU Vitamin D3 | Placebo
Started | 31 | 31
Completed | 30 | 31
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Postmenopausal women with 25(OH)D 10 - 29 ng/ml.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2000 IU Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.7) | 65.9 (8.2) | 67.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum 25-hydroxy Vitamin D3
Description: Our primary outcome variable is the effect of supplementation on change in serum 25(OH)D3;
Time Frame: Baseline, 1 and 4 months post supplementation
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 2000 IU Vitamin D3 | Placebo
Number analyzed (Participants) | 30 | 31
ng/ml
  One Month | 6.0 (4.1) | -0.8 (4.3)
  Four Month | 10.4 (5.8) | 0.3 (4.1)

2. Secondary Outcome: Change in Parameters of the Vitamin D Assay Panel
Description: Secondary outcomes are change in cholecalciferol, 24,25(OH)D3 and free 25(OH)D3.
Time Frame: Baseline, 1 and 4 months post supplementation
Population: Postmenopausal Caucasian women with 25(OH)D < 10 > 30 ng/ml
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 2000 IU Vitamin D3 | Placebo
Number analyzed (Participants) | 30 | 31
ng/ml
  Cholecalciferol Month 1 | 6.7 (4.3) | -0.6 (1.3)
  Cholecalciferol Month 4 | 6.7 (5.7) | -0.20 (2.12)
  24,25(OH)D3 Month 1 | 0.3 (.08) | -0.2 (0.5)
  24,25(OH)D3 Month 4 | 1.2 (0.91) | -0.1 (0.56)
  free 25(OH)D3 Month 1 | 1.3 (1.3) | -0.2 (1.0)
  free 25(OH)D3 Month 4 | 2.4 (1.9) | -0.1 (1.3)

ADVERSE EVENTS:
Time Frame: From screening to 4m visit, period covered ~6m
Arm/Group | 2000 IU Vitamin D3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 4/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2000 IU Vitamin D3 (N=31) | Placebo (N=31)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) — Two subjects noted experiencing diarrhea over the study course.
Depression (Psychiatric disorders) | 0 (0) | 2 (2) — Two subjects reported a new diagnosis of depression and starting pharmaceutical intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No